CLINICAL TRIAL: NCT04924413
Title: L-TIL Plus Tislelizumab as First-line Treatment in Advanced Malignant Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Quanli Gao (Other Government)
Responsible Party: Sponsor-Investigator, Quanli Gao, Head of Immunotherapy, Henan Cancer Hospital
Organization: Henan Cancer Hospital (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HenanCH L-TIL Melanoma
Record Dates: First submitted 2021-05-31; First posted 2021-06-14 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — tislelizumab

STUDY DESIGN:
Intervention Model Description: L-TIL and Tislelizumab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- L-TIL and Tislelizumab (Experimental): L-TIL（3-10）x10*9/m2, Q3W, 4 cycles Tislelizumab 200mg, iv, Q3W, 1 year
  Interventions: Drug: Tislelizumab

INTERVENTIONS:
Drug: Tislelizumab — PD-1 positive lymphocytes are isolated from peripheral blood and amplified for transfusion
  Other Names: L-TIL

SUMMARY:
The main purpose of this study is to evaluate the safety and effectiveness of liquid tumor infiltrating lymphocytes (L-TIL) combined with tislelizumab as the first-line treatment in patients with advanced malignant melanoma. This study plan to include stage III or IV unresectable or metastatic cutaneous or acral malignant melanoma patients, treat with L-TIL 4 cycles with each infusion (3 -10) x10*9/m2 cells, combined with tislelizumab 200mg, iv, Q3W. It is expected that 30 patients will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological confirmed melanoma 2. Advanced stage confirmed by radiological examination 3. Untreated 4. ECOG PS 0-1 6. Good organ function 7. No other severe diseases such as autoimmune disease, organ transplant, chronic infection.

8. Other tumor disease.

Exclusion Criteria:

1. Symptomatic brain metastases
2. Active infection
3. Active HBV or HCV infection
4. HIV infection
5. Autoimmune disease
6. Sensitive to drug or ingredients
7. Severe mental disorders
8. Sever disfunction of heart, liver and kidney

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-07-02 (Actual)

PRIMARY OUTCOMES:
Efficacy (ORR) | 8 weeks
  The objective response rate (ORR) at 8 weeks from baseline.
Efficacy (ORR) | 16 weeks
  The objective response rate (ORR) at 16 weeks.
Efficacy (DOR) | 1 year
  The duration of response (DOR) at 1-year.
Efficacy (DOR) | 2 years
  The duration of response (DOR) at 2-year.

SECONDARY OUTCOMES:
Progression free survival (PFS) | 1 year
  The PFS rate at 1 year.
Progression free survival (PFS) | 2 years
  The PFS rate at 2-year.
Overall survival (OS) | 1 year
  The OS rate at 1 year.
Overall survival (OS) | 2 years
  The OS rate at 2-year.
Safety (adverse events) | 2 years
  The adverse events followed by treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Quanli Gao, Ph.D, Study Director — Henan Cancer Hospital
Locations (1):
- Affiliated Cancer Hospital of Zhengzhou University & Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li T, Zhao L, Yang Y, Wang Y, Zhang Y, Guo J, Chen G, Qin P, Xu B, Ma B, Zhang F, Shang Y, Li Q, Zhang K, Yuan D, Feng C, Ma Y, Liu Z, Tian Z, Li H, Wang S, Gao Q. T Cells Expanded from PD-1+ Peripheral Blood Lymphocytes Share More Clones with Paired Tumor-Infiltrating Lymphocytes. Cancer Res. 2021 Apr 15;81(8):2184-2194. doi: 10.1158/0008-5472.CAN-20-2300. Epub 2021 Jan 6. PMID 33408117